CLINICAL TRIAL: NCT01485744
Title: A Phase 1b Clinical Trial of LDE225 in Combination With Fluorouracil, Leucovorin, Oxaliplatin and Irinotecan (FOLFIRINOX) in Previously Untreated Locally Advanced or Metastatic Pancreatic Adenocarcinoma, With an Expansion Cohort at the Recommended Phase 2 Dose
Brief Title: LDE225 With Fluorouracil, Leucovorin, Oxaliplatin, and Irinotecan for Untreated Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Jeffrey W. Clark, MD, Physician Hematology/Oncology, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-164
Record Dates: First submitted 2011-12-01; First posted 2011-12-05 (Estimated); Last update posted 2020-08-04 (Actual); Status verified 2020-07

CONDITIONS: Pancreatic Cancer
Keywords: metastatic; untreated; advanced
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasm Metastasis | interventions — sonidegib; Fluorouracil; Leucovorin; Oxaliplatin; Irinotecan; folfirinox

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- LDE225; Fluorouracil; Leucovorin; Oxaliplatin; Irinotecan (Experimental)
  Interventions: Drug: LDE225; Fluorouracil; Leucovorin; Oxaliplatin; Irinotecan

INTERVENTIONS:
Drug: LDE225; Fluorouracil; Leucovorin; Oxaliplatin; Irinotecan — LDE225 200-800 mg daily orally. Fluorouracil 2400 mg IV every other week. Irinotecan 180 mg/m2 IV every other week. Oxaliplatin 85 mg/m2 IV every other week. Leucovorin 400 mg/m2 IV every other week.
  Other Names: FOLFIRINOX; 5-FU; CPT-11

SUMMARY:
LDE225 is a new medicine that blocks the Hedgehog (Hh) pathway. The Hh pathway is a cascade of molecular events that control cell growth and have been linked with the development of many human cancers, including pancreatic cancer. Information from research studies suggests that LDE225 in combination with FOLFIRINOX may help to stop the growth of cancer cells. In this research study, the investigators are looking to determine the maximum dose of LDE225 in combination that can be given safely to patients with locally advanced or metastatic pancreatic cancer.

DETAILED DESCRIPTION:
Study medication will be given in cycles of 14 days. Subjects will keep a study drug diary for each treatment cycle. LDE225 capsules will be taken by mouth in the morning every day of each cycle.

On days 1-2 of each cycle, subjects will take LDE225 at the clinic followed by FOLFIRINOX intravenous infusion (through a vein).

Subjects will come to the clinic weekly for the first 5 weeks, then every other week (Week 7, 9, 11, etc.) and receive the following procedures:

Review of current medications and any side effects Physical exam Performance Status Blood tests (2 teaspoons of blood) Assessment of tumor (repeated every 8 weeks) ECG at week 3 and 5

Subjects will also have pharmacokinetic (PK) blood samples taken. PK samples are used to find out the amount of study medication in the blood. Each PK sample is about 1/2 teaspoon of blood. Subjects will have PK samples taken on:

Day 1 of Cycles 1, 2, 3, 4, 6, and 7 before the dose of LDE225 Day 1 of Cycle 5 - drawn before the first dose of LDE225 and at 1, 2, 3, 4, 5, and 6 hours Day 2 of Cycle 5: One PK blood sample

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed locally advanced or metastatic pancreatic adenocarcinoma
* Previously untreated locally advanced or metastatic pancreatic adenocarcinoma. Pts newly diagnosed with metastatic recurrence after adjuvant therapy for resected disease are eligible, if completion of adjuvant therapy was > 8 months ago
* Measurable disease
* Adequate organ and marrow function
* Able to take oral drugs

Exclusion Criteria:

* Concurrent active primary or metastatic cancer other than superficial squamous cell or basal cell skin cancer
* Pregnant or breastfeeding
* Receiving any other standard or investigation anticancer agents, with the exception of hormonal therapy
* Prior chemoradiation to the primary pancreatic tumor unless there is a measurable distant site of disease
* Known CNS metastases
* History of hypersensitivity reactions to any components of the treatment regimen
* Known malabsorption syndromes
* Neuromuscular disorders
* Receiving other anti-neoplastic therapy concurrently
* Requires warfarin/Coumadin for therapeutic coagulation
* Receiving treatment with medications known to be moderate and strong inhibitors or inducers of CYP3A4/5
* Uncontrolled diarrhea
* Peripheral neuropathy > grade 1 due to any cause
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia other than chronic atrial fibrillation, or psychiatric illness/social situations that would limit compliance with study requirements
* HIV positive

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2011-12; Primary Completion 2019-11 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | 2 years
  To determine the maximal tolerated doses of LDE225 in combination with FOLFIRINOX in patients with locally advanced or metastatic pancreatic adenocarcinoma
Toxicity | 2 years
  To determine the types, frequency, and severity of adverse events occurring in subjects receiving LDE225 in combination with FOLFIRINOX

SECONDARY OUTCOMES:
Response Rate | 2 years
  To determine the response rate of pancreatic cancers treated with LDE225 in combination with FOLFIRINOX

CONTACTS AND LOCATIONS:
Overall Officials: Jeffery W Clark, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts